CLINICAL TRIAL: NCT05518383
Title: B-cell Mature Non-Hodgkin's Lymphoma Treatment Protocol in Children and Adolescents 2021 (B-NHL-M-2021)
Brief Title: B-cell Mature Non-Hodgkin's Lymphoma Treatment Protocol in Children and Adolescents 2021
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2021-07
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-05

CONDITIONS: Non-hodgkin Lymphoma,B Cell; Burkitt Lymphoma; Primary Mediastinal Lymphoma; Primary CNS Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: B-cell mature non-Hodgkin's lymphoma; Burkitt's lymphoma; Diffuse large B-cell lymphoma; primary mediastinal lymphoma, primary CNS lymphoma; rituximab; children, adolescents; treatment
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Ifosfamide; Methotrexate; Vincristine; Doxorubicin; Lomustine; Carmustine; Melphalan; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R1: stage I and II (Experimental): R1: resection status: complete, stage I and II
  Interventions: Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Etoposide, Ifosfamide, Methotrexate
- R2: incomplete, stage I and II (Experimental): R2: resection status: incomplete, stage I and II
  Interventions: Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Etoposide, Ifosfamide, Methotrexate, Vincristine
- R3: incomplete, stage III and LDH < 2 x ULN (Experimental): R3: resection status: incomplete, stage III and LDH < 2 x ULN
  Interventions: Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Doxorubicin hydrochloride, Etoposide, Ifosfamide, Methotrexate, vincristine
- R4: stage III and LDH ≥ 2 x ULN, stage IV/B-AL and CNS negative; CNS + (Experimental): R4: resection status: incomplete, stage III and LDH ≥ 2 x ULN, stage IV/B-AL and CNS negative; CNS +
  Interventions: Drug: Cyclophosphamide , Cytarabine, Dexamethasone, Doxorubicin hydrochloride, Etoposide, Ifosfamide, Methotrexate, Vincristine, Сarboplatine, CCNU/ BCNU, Melphalan, Idarubicin

INTERVENTIONS:
Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Etoposide, Ifosfamide, Methotrexate — For patients with very limited disease (R1- stage I/II СR), the addition of rituximab might allow the omission of anthracyclines and vincristine without jeopardizing survival rates but reducing acute and long term toxicities. In this treatment arm, it is tested whether the event-free survival is similar to that of the historical control
  Arms: R1: stage I and II
Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Etoposide, Ifosfamide, Methotrexate, Vincristine — R2: Drug: Rituximab 2 doses of Rituximab (375 mg/m²) before the start of the first chemotherapy cycle, 2 doses of Rituximab before the start of the second chemotherapy cycle
  Arms: R2: incomplete, stage I and II
Drug: Cyclophosphamide, Cytarabine, Dexamethasone, Doxorubicin hydrochloride, Etoposide, Ifosfamide, Methotrexate, vincristine — 2 doses of Rituximab (375 mg/m²) before the start of the first chemotherapy cycle, 2 doses of Rituximab before the start of the second
  Arms: R3: incomplete, stage III and LDH < 2 x ULN
Drug: Cyclophosphamide , Cytarabine, Dexamethasone, Doxorubicin hydrochloride, Etoposide, Ifosfamide, Methotrexate, Vincristine, Сarboplatine, CCNU/ BCNU, Melphalan, Idarubicin — Rituximab 4 doses of Rituximab (375 mg/m²) before the start of the first chemotherapy cycle, Further
  Arms: R4: stage III and LDH ≥ 2 x ULN, stage IV/B-AL and CNS negative; CNS +

SUMMARY:
The aim of the trial is to evaluate the molecular characteristics and MDD/MRD of B-NHL in pediatric patients in order to identify on the one hand the very high risk group and to prescribe them more intensive treatment on the other hand to identify those patients who don't need very aggressive therapy. One more study question is to evaluate the role of PET/CT in assessment of the completeness of remission.

The following primary study questions are going to be analyzed:

* the effectiveness (event-free survival) in pediatric patients with very limited mature B-NHL (R1 - stage I and II R) of substituting anthracyclines and vincristine by the rituximab without compromising survival rates.
* the effectiveness (event-free survival) in pediatric patients with limited mature B-NHL (R2 - stage I and II NR) of substituting anthracyclines by the rituximab without compromising survival rates.
* the effectiveness (event-free survival) in pediatric patients with advanced VHR mature B-NHL (R4 - stages with unfavourable genetics of substituting standard chemotherapy by "second-line" block VICI in order to improve results

Secondary study questions will address

* additional parameters for immune reconstitution, lymphocyte subpopulations, immunoglobulin levels, vaccination titers and infection rates
* kinetics of immune reconstitution after treatment

DETAILED DESCRIPTION:
Detailed Description:

Risk group stratification:

R1: resection status: complete, stage I and II R2: resection status: incomplete, stage I and II R3: resection status: incomplete, stage III and LDH < 2 x ULN R4: resection status: incomplete, stage III and LDH ≥ 2 x ULN, stage IV/B-AL and CNS negative; CNS +

For patients with very limited disease (R1- stage I/II СR), the addition of rituximab might allow the omission of anthracyclines and vincristine without jeopardizing survival rates but reducing acute and long term toxicities. In this treatment arm, it is tested whether the event-free survival is similar to that of the historical control For patients with limited disease (R2- stage I/II NR), the addition of rituximab might allow the omission of anthracyclines without jeopardizing survival rates but reducing acute and long term toxicities.

For patients with limited disease (R3 - stage III and LDH < 2 x ULN ), the addition of rituximab might allow reduce the number of blocks to four without jeopardizing survival rates but reducing toxicities For patients with obligate factors of poor prognosis (additional adverse cytogenetic findings (TP-53, 11qLOH) it is tested whether the event-free survival can be improved by adding rituximab and adding blocks R-VICI

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis 0 to 18 years.
* The diagnosis of Burkitt's lymphoma, Diffuse large B-cell lymphom, primary mediastinal lymphoma, primary CNS lymphoma, B-cell (Burkitt) AL
* Informed consent of the patient parents (guardians) to be treated

Exclusion Criteria:

* previous malignancy, prior organ transplant, HIV infection or AIDS or severe immunodeficiency
* hypersensitivity to rituximab or to ingredients of other IMPs.
* no informed consent of the patient parents (guardians) to be treated

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years after the start of therapy
  Event-free survival The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies.
Event-free survival | 7 years after the start of therapy
  Event-free survival The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies.

SECONDARY OUTCOMES:
assessment of MDD and MRD indicators, p53 and 11qLOH status in patients on the B-NHL-M-2021 protocol | 3 years after the start of therapy
assessment of MDD and MRD indicators, p53 and 11qLOH status in patients on the B-NHL-M-2021 protocol | 7 years after the start of therapy
assessment of PET-CT results - initial and control points (early PET response).after the 2nd block | after the 2nd block - CT with CL of the involved areas, PET-CT examination on the 14th day (maximum on the 17th day) after the last injection of CT, IPT, MRD in the bone marrow - after 4th block - CT with the CL of the involved areas
  measurement of tumor volume at diagnosis and measurement of tumor volume reduction after therapy in percent after the 2nd block - CT with CL of the involved areas, PET-CT examination on the 14th day (maximum on the 17th day) after the last injection of CT, IPT, MRD in the bone marrow
assessment of PET-CT results - initial and control points (early PET response) after 4th block | PET-CT examination on the 14th day (maximum on the 17th day) after the last administration of CT, MRD in the bone marrow if present after the 2nd block
  measurement of tumor volume at diagnosis and measurement of tumor volume reduction after therapy in percent after 4th block - CT with the CL of the involved areas , PET-CT examination on the 14th day (maximum on the 17th day) after the last administration of CT, MRD in the bone marrow if present after the 2nd block After the 6th block - CT with CL of the involved areas
Relapse-free survival (RFS) | 3 years after the start of therapy
  RFS is defined as time from start of treatment up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Relapse-free survival (RFS) | 7 years after the start of therapy
  RFS is defined as time from start of treatment up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Response rate (RR) [ and after second course and after two injections of rituximab]. Complete response, partial remission, stable disease or progressive disease | 3 years after the start of therapy
Response rate (RR) [ and after second course and after two injections of rituximab]. Complete response, partial remission, stable disease or progressive disease | 7 years after the start of therapy
Rate of patients achieving normal immunoglobulin level | 12 months after start of treatment
Rate of patients with normal lymphocyte subpopulations in the peripheral blood 12 months after start of treatment | 12 months after start of treatment
Interval to normal lymphocyte subpopulations in the peripheral blood. | 7 years after the start of therapy
Rate of patients with sufficient titers after vaccination one year after start of treatment | 1 year after start of treatment
Immune reconstitution rate (only in R1/R2 patients) | 1 year after start of treatment
Time interval from start of treatment to normal CD19 positive B-cells in the peripheral blood. | 1 year after start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, RF, Russia